CLINICAL TRIAL: NCT06096272
Title: A Pilot Study Using Exergaming With Augmented Reality to Promote Physical Activity in Children With Cerebral Palsy
Brief Title: Using Augmented Reality to Promote Physical Activity in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Melissa Bent, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-23-00120
Record Dates: First submitted 2023-08-28; First posted 2023-10-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy; Mobile Phone Use; Pediatric ALL; Physical Disability; Physical Inactivity
MeSH Terms: conditions — Cerebral Palsy; Cell Phone Use; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augment Therapy app (Experimental): The app will be implemented with the participant's compatible iPad that will be securely integrated with a network-server for real-time data access and storage. If the participant does not have a compatible device, this will be provided by the research team. Participants will be provided an on-site or virtual CHLA tutorial about using the app and set up of the gaming system. Participants will access their home program on the app at least for 20 minutes, 3 times a week over a 4-week period. A coordinator will check in virtually with the participant during the program. They will complete baseline and final surveys. Exercise data will be collected and stored through the Augment Therapy™ app and self log book.
  Interventions: Device: Augment Reality Exergames

INTERVENTIONS:
Device: Augment Reality Exergames — Adaptive physical activity AR gaming modules were created in collaboration with physical therapists with expertise in CP and the Augment Therapy app development team. The program will consists of 5 games adapted for children with cerebral palsy.

SUMMARY:
Children with cerebral palsy (CP), Gross Motor Functional Classification Scale (GMFCS) I-II will be recruited to participate in a home based physical activity intervention for 4 weeks. Demographic data will be collected, and validated surveys assessing baseline physical activity level and mobility will be completed. Participants will have an exercise program assigned and will be given a logbook to record their exercise adherence. They will be assigned to the Augment Reality (AR) app group. The AR app group will have exercises administered through the AR app. At the end of the program, participants will complete final surveys and an exit interview.

DETAILED DESCRIPTION:
Muscle weakness in cerebral palsy (CP) results in a reduced level of physical activity. Reduced physical activity can lead to adverse health consequences. Augmented reality (AR) is increasingly being used to promote physical activity. The purpose of this study is to determine if adaptive exercise gaming program utilizing AR mobile app for children with cerebral palsy can promote physical activity through a prospective pilot study.

Children with CP, GMFCS I-II between the ages of 5-18 years old will be recruited to participate in a home-based physical activity AR games.

Study Population: Inclusion criteria are: diagnosis of cerebral palsy, ambulatory (GMFCS I and II), ages 5-18 years, English or Spanish speaking, and no plans for lower extremity surgery in the next 2 months. Exclusion criteria are: moderate to severe developmental or cognitive delay, severe visual or hearing condition, recent casting or surgical procedure over the past 4 months that impacts physical activity, or G-tube dependent. Interested participants will be scheduled for a virtual or in person visit in which informed consent will be obtained.

Study Design: All participants will use the app for 4-weeks. The app will be implemented with an iPad® provided by the research team if the participant does not have a compatible device, that will be securely integrated with a network-server for real-time data access and storage. Participants will be provided an on-site or virtual CHLA tutorial about using the app and set up of the gaming system. Augment Therapy support personnel will assist with home set up if needed. Participants will access their home program on the app at least for 20 minutes, 3 times a week over a 4-week period. A coordinator will check in virtually with the participant during the course of the program. Exercise data will be collected and stored through the Augment Therapy™ app and self log book. Feasibility will be defined as 1) Program Engagement measured by the app and program evaluation surveys 2) Program Adherence measured by exercise compliance defined as the number of self-reported exercises logged, app usage logs, and sessions completed for the intervention and control groups. Validated questionnaires will be administered to evaluate the effect of the intervention at baseline and final assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy,
* Ambulatory (GMFCS I and II)
* English or Spanish speaking
* No plans for lower extremity surgery in the next 4 months

Exclusion Criteria:

* Moderate to severe developmental or cognitive delay
* Significant hearing loss or visual impairment
* Recent surgical procedure or fracture over the past 4 months that impacts physical activity

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that complete mobile application delivered exercise program. | Baseline to 4 weeks.
  Measured by proportion of time in the mobile application (180/360 total minutes).
Number of participants that complete the standard exercise program. | Baseline to 4 weeks.
  Measured by proportion of time (180/360 total minutes) to complete exercises in logbook.

SECONDARY OUTCOMES:
Engagement in the mobile application, Gold-Rizzo Immersion and Presence (GRIP) Inventory scale. | At Week 4.
  Measured by the Gold-Rizzo Immersion and Presence (GRIP) Inventory scores in the domains of immersion, feasibility, realism, transportation and satisfaction, higher scores reflect better experience.
Change in Quality-of-Life measure: Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Activity and Mobility. | Baseline to 4 weeks.
  Measure at baseline and end of intervention, change of PROMIS Physical Activity and Mobility scores, higher scores represent higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bent, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Jackie and Gene Autry Orthopedic Center, CHLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No